CLINICAL TRIAL: NCT07018921
Title: Do Sweeteners Need to be Tasted to Affect Appetite? A Pilot Study
Brief Title: Low Calorie Sweeteners Effects on Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Nikoleta Stamataki, Dr Nikoleta Stamataki, University of Manchester
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2022-15284-25905
Record Dates: First submitted 2023-03-16; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2023-03

CONDITIONS: Appetite
MeSH Terms: interventions — rebaudioside A

STUDY DESIGN:
Intervention Model Description: This study is double blind. All participants are completing 2 testing sessions in randomised and counterbalanced order. Participants and researchers (who are also outcome assessors) are blinded to the beverages content. Un-blinding will be performed following analysis of results.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will attend 2 testing sessions, where they will consume either the stevia capsule or the placebo capsule in a double-blind randomised crossover design.
  Interventions: Dietary Supplement: rebaudioside A; Dietary Supplement: Placebo
- rebaudioside A (Active Comparator): Participants will attend 2 testing sessions, where they will consume either the stevia capsule or the placebo capsule in a double-blind randomised crossover design.
  Interventions: Dietary Supplement: rebaudioside A; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: rebaudioside A — rebaudioside A encapsulated in a vegetarian capsule
Dietary Supplement: Placebo — carboxymethylcellulose encapsulated in a vegetarian capsule

SUMMARY:
The principal research question is whether the ingestion of stevia (rebaudioside A) in encapsulated format will have any effects on blood glucose, appetite and food intake in healthy human volunteers.

DETAILED DESCRIPTION:
Obesity presents a major global health crisis; developing healthier diets is a key goal. Excess consumption of caloric sweeteners contributes to the alarming high rates of overweight and obesity. Non-nutritive sweeteners, like stevia, are used to decrease energy content of foods and beverages. Very recently a systematic review and meta-analysis conducted and published by WHO, concluded that non-nutritive sweeteners use results in small reduction in body weight and BMI in adults, as assessed in RCTs.

In a previous set of studies from our group we showed that a single-dose of a stevia-sweetened beverage prior to lunch leads a lower energy intake compared to consuming water or a sugar-sweetened beverage (Stamataki et al J Nutr. 2020; 150(5):1126-1134. doi: 10.1093/jn/nxaa038). This effect was confirmed to be present in the long-term, as in another 12-weeks trial we demonstrated that individuals in the stevia group (they started consuming stevia drops twice daily with habitual drinks before their meals) demonstrated a significant spontaneous reduction in energy intake compared to the control group (Stamataki et al Nutrients. 2020;12(10):3049. doi: 10.3390/nu12103049).

In a nutshell, this research so far has showed that stevia consumption elicits benefits in appetite and energy intake, without affecting physiological responses such as postprandial glucose response. Taking this research a step further, it is crucial now to answer whether sweetness without calories was the key component of these outcomes, in other words would stevia have the same effects if it was not tasted, if sweet taste (in the oral cavity) was bypassed?

As such the main aim of this study is to evaluate the effects of stevia in a capsule vs placebo on appetite and energy intake and elucidate whether stevia elicits similar effects when sweet taste is bypassed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 40 years
* BMI between 18.5-24.9 kg/m2
* DEBQ for restraint eating ≤ 3
* Healthy - general good health
* Currently not taking any medication (other than females taking the oral contraceptives, or medication that does not affect taste, and glucose response)
* Regular breakfast eaters (≥5 times per week)
* Stable weight, ≤ 5 kg last 3 months
* No self-reported food allergy or intolerance to foods supplied during the study
* The participant is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The participant is able to read, comprehend and record information written in English.
* A signed and dated written informed consent is obtained from the participant.

Exclusion Criteria:

* Age under 18 years or over 40 years old.
* BMI ≥25 kg/m2 and <18.5kg/m2
* Subjects who are currently on a diet
* Subjects who follow special diets for weight maintenance, such as Atkins Diet, Weight Watchers, gluten-free diet, The Zone diet, Raw Food Diet etc.
* Vegetarians, vegans
* Subjects having breakfast fewer than 5 times per week.
* Presence of any chronic condition requiring medication that might affect our results (e.g. diabetes, mental diseases, gastrointestinal diseases)
* Subjects with eating disorders (binge eating disorder, bulimia etc)
* Subjects who are currently experiencing anxiety or depression.
* Participants who drink more than the NHS guidelines (14 units per week)
* Participants who are, or may be, pregnant, or currently lactating.
* Subjects who regularly consume dietary supplements for weight loss, muscle building etc.
* Subjects who have aversions to foods related with the study.
* Subjects with food allergies or intolerance related with the foods/ drinks of the study.
* Habitual NNS consumers, >1 can of diet beverage or >1 sachet of low calorie sweeteners (corresponding to 1 spoonful) per week.
* The participant cannot read, comprehend and record information written in English.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Energy intake | Lunch at 30 min after the ingestion of the treatment
  Participants are allowed to eat from a buffet lunch until they feel comfortably full.

SECONDARY OUTCOMES:
Appetite ratings | 0, 15, 30 and 60 min
  Using VAS scales for appetite, participants rate their appetite at baseline (before ingestion of the capsule), 15, 30 min after the ingestion of the capsule as well as at 60 min (which also corresponds 30 min after the start of the ad libitum meal).
Blood glucose | 0, 15, 30 and 60 min
  Capillary blood glucose measurements will be conducted at baseline (0), 15 min and 30 min following treatment as well as at 60 min after the ingestion of the capsule which also corresponds 30 min after the consumption of the ad libitum lunch.

OTHER OUTCOMES:
Meal attributes in VAS scales | 60 min
  pleasantness, sweetness, saltiness and familiarity of the buffet meal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided